CLINICAL TRIAL: NCT07356024
Title: Effect of Acupressure on Blood Glucose And Anxiety in Elderly With Diabetes: A Three Arm, Parallel Group, Double Blind, A Randomized Controlled Trial
Brief Title: Effect of Acupressure on Blood Glucose And Anxiety in Elderly With Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Saadet Can Çiçek, Associate Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BAIBU-SBF-YO-2025
Record Dates: First submitted 2026-01-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus; Acupressure
Keywords: Randomized Controlled Trial; Diabetes; Elderly; Acupressure; Anxiety; Blood Glucose
MeSH Terms: conditions — Diabetes Mellitus; Anxiety Disorders | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three parallel groups: an acupressure intervention group, a sham acupressure (placebo) group, or a control group receiving routine care.
Who Masked: Participant, Outcomes Assessor
Masking Description: Data collection and data entry will be performed by trained personnel independent of the intervention process. All data will be recorded and entered into the dataset using coded identifiers only. Participants will be blinded to group allocation, and the statistician performing the data analysis will also be blinded to group assignments. The study will therefore be conducted using a double-blind design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure Group (Experimental): Participants assigned to this group will receive acupressure applied to the HT7, SP6, and ST36 acupoints by a trained researcher. The intervention will be administered once daily for six sessions, with each session lasting approximately 15-20 minutes, in addition to routine clinical care.
  Interventions: Other: Acupressure
- Placebo Group (Placebo Comparator): Participants assigned to this group will receive sham acupressure, consisting of light pressure applied to non-acupoint areas near the same anatomical regions as the intervention group. The sham procedure will be administered once daily for six sessions, with each session lasting approximately 15-20 minutes, in addition to routine clinical care. Pressure will be applied on the bone area where the meridians do not pass, parallel to the points where acupressure is applied to the sham points (approximately 1-1.5 cm away).
  Interventions: Other: Placebo Sham Acupressure
- Control Group (Routine Care) (Other): Participants assigned to this group will receive routine clinical care only and will not receive any additional intervention during the study period.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Acupressure — The acupressure intervention will be conducted in a designated room at the institution, once daily for 6 consecutive days, with each session lasting 15-20 minutes, totaling 6 sessions. During the first 3-5 minutes of each session, participants will be guided to the appropriate position and approached to ensure comfort. Acupressure will then be applied to a total of six points: both wrists (HT7) and both legs (ST36, SP6), with two points on each limb. Each of the six points will receive a 30-second preparation followed by 2 minutes of acupressure application
  Arms: Acupressure Group
Other: Placebo Sham Acupressure — Participants in the placebo group will receive sham acupressure administered by the researcher in a quiet, designated room at the institution, once daily for 6 consecutive days, with each session lasting 15-20 minutes, totaling 6 sessions. Pressure will be applied to bony areas approximately 1.5-2 cm away from the HT7, SP6, and ST36 points, where no meridians pass. Prior to the application, the sham points will be gently warmed and massaged for approximately 20 seconds to reduce tissue sensitivity, preparing the area for the sham acupressure procedure.
  In the intervention group, evaluation will be made at the specified frequency, using the same measurement tools and the same measurement methods.
  Arms: Placebo Group
Other: Routine care — Participants will receive routine clinical care only and no additional intervention.
  Arms: Control Group (Routine Care)

SUMMARY:
This study is designed to evaluate the effect of acupressure on blood glucose levels and anxiety in elderly individuals with diabetes. Participants will be assigned to an acupressure intervention group or a control group. The primary outcome of the study is blood glucose level, which will be assessed at baseline and at the end of the intervention period. Secondary outcomes include anxiety levels.

DETAILED DESCRIPTION:
This study is a prospective, interventional, randomized, double-blind, controlled trial designed to evaluate the effect of acupressure on blood glucose levels and anxiety in elderly individuals with diabetes. Eligible participants will be randomly assigned to one of three groups: an acupressure intervention group, a sham acupressure (placebo) group, or a control group receiving routine care.

Participants in the intervention group will receive acupressure applied to the HT7, SP6, and ST36 acupoints by a trained researcher. The intervention will be administered once daily for six sessions, with each session lasting approximately 15-20 minutes. The sham acupressure group will receive light pressure applied to non-acupoint areas near the same anatomical regions, while the control group will continue to receive routine clinical care without any additional intervention.

The primary outcome of the study is blood glucose level, assessed using fasting and postprandial capillary blood glucose measurements at baseline and at predefined time points during the intervention period. Secondary outcomes include anxiety levels, measured using the State-Trait Anxiety Inventory. Outcome assessments will be conducted by assessors blinded to group allocation.

Prior to the main trial, a pilot study will be conducted to evaluate the feasibility of the intervention protocol and data collection procedures, and to estimate the effect size required for calculating the final sample size of the main study. Findings from the pilot study will be used to refine the intervention procedures and to determine the final sample size. Participants included in the pilot study will not be included in the main trial.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreeing to participate in the study,
* Being 65 years of age or older,
* Having been diagnosed with diabetes for at least one year,
* Not having any hearing, speech, or vision impairments that would interfere with communication,
* Being able to speak and understand Turkish,
* Having a Mini-Mental State Examination (MMSE) score of 23 or higher for literate participants and 19 or higher for illiterate participants,
* Not using any other complementary or supportive therapies during the study period,
* Receiving dietary treatment or oral antidiabetic medication for diabetes management,
* Having no skin irritation, ulceration, or other impairment of skin integrity at the application sites.

Exclusion Criteria:

* Initiation of a new medication with potential effects on blood glucose levels in addition to the current treatment during the study period,
* Use of insulin therapy for diabetes management.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-24 (Estimated); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-10-27 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose | Baseline to Day 6
  Participant's blood glucose results will be evaluated by capillary blood glucose measurement after at least 8-10 hours of fasting and 2 hours after meals in a postprandial state.
  Measurement Process:
  Fasting blood sugar measurement: Fasting blood glucose will be evaluated before starting the application, after 3 sessions and 24 hours after the end of 6 sessions, after an 8-10 hour fast.
  Postprandial blood glucose measurement: Postprandial blood glucose levels will be assessed at the 2nd hour after the first bite of the meal. The first postprandial blood glucose assessment will take into account the first meal after the first session, the second assessment will take into account the first meal after the 3rd session, and the third assessment will take into account the postprandial blood glucose levels measured at the first meal after the 6th session.
Anxiety | Baseline to Day 6
  Anxiety levels will be assessed using the Spielberger State-Trait Anxiety Inventory (STAI). The Spielberger State-Trait Anxiety Inventory (STAI) is a validated self-report questionnaire used to assess anxiety. It consists of two distinct subscales:
  State Anxiety (STAI-S), which measures temporary anxiety related to the individual's current condition, and Trait Anxiety (STAI-T), which measures a person's general and long-term tendency to experience anxiety.
  Each subscale includes 20 items, with total scores ranging from 20 to 80. Higher scores indicate higher levels of anxiety, while lower scores indicate lower anxiety levels.
  Measurement Process:
  Before the intervention, the Spielberger State-Trait Anxiety Inventory (STAI) will be administered. The Spielberger State Anxiety Inventory will be applied to the participants half an hour after the first session, before the sixth session, and half an hour after the completion of the sixth session to assess their current anxiety levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No